CLINICAL TRIAL: NCT01955421
Title: A Randomized, Open-label Phase II Trial of Erlotinib 100mg Daily Versus Gefitinib 250mg Daily in Patients With Advanced Non-small Cell Lung Cancer Who Harbor EGFR Mutations.
Brief Title: Erlotinib 100mg qd Versus Gefitinib 250mg qd for EGFR Mutant Nsclc
Acronym: NSCLC EGFR TKI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E100VG250; Tarceva100vsIressa250 (Registry Identifier: Tarceva100vsIressa250)
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Advanced Stage Non Small Cell Lung Cancer
Keywords: NSCLC; stage IIIB; stage IV); confirmed by histology or cytology methods; Harboring a PCR-confirmed activating mutation of EGFR, including an exon 19 deletion or an exon 21 L858R point mutation
MeSH Terms: interventions — Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib100 (Experimental): Patients will be randomized to buy and receive erlotinib 100mg qd.
  Interventions: Drug: Erlotinib 100mg qd
- Gefitinib250 (Experimental): Patients will be randomized to buy and receive gefitinib 250mg qd.
  Interventions: Drug: Gefitinib 250mg qd

INTERVENTIONS:
Drug: Erlotinib 100mg qd
  Arms: Erlotinib100
Drug: Gefitinib 250mg qd
  Arms: Gefitinib250

SUMMARY:
This study is a multicenter, randomized, open-label Phase II trial that compares reduced dose erlotinib 100mg daily and standard dose gefitinib 250mg daily in patients with advanced non-small cell lung cancer who harbor EGFR mutations. The primary endpoint is disease control rate (DCR) and the key secondary endpoint is progression free survival (PFS). A total of 224 eligible patients will be randomized to receive either erlotinib 100mg daily or gefitinib 250mg daily in a 1:1 ratio until patients experience disease progression. Independent assessment of the major endpoints will be completed in a treatment-blinded manner. Randomization will be stratified based on treatment-lines (first-line vs. maintenance vs. second-line therapy). Tumor response and progression will be assessed according to RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced stage NSCLC (stage IIIB or IV) which is confirmed by histology or cytology methods.
2. Harboring a PCR-confirmed activating mutation of EGFR, including an exon 19 deletion or an exon 21 L858R point mutation.
3. Measurable disease according to RECIST1.1.
4. Eastern Cooperative Oncology Group (ECOG) score of 0-2
5. Adequate organ function, defined as all of the following:

   1. LVEF >50% or within institution normal values.
   2. Absolute neutrophil count (ANC)>1500/mm3.
   3. Platelet count >75,000/mm3
   4. Estimated creatinine clearance>45m1/min.
   5. Total bilirubin<1.5 times institutional ULN (Patients with Gilbert's Syndrome total bilirubin must be <4 times institutional ULN).
   6. Aspartate amino transferase (AST) or alanine amino transferase (ALT) < three times the institutional upper limit of normal (ULN) (if related to liver metastases<five times institutional ULN).
6. Recovered from any previous therapy related toxicity to ≤CTCAE Grade 1 at study entry (except for stable sensory neurupethy ≤CTCAE Grade 2 and alopecia).
7. Ability to take oral medication in the opinion of the investigator.
8. Age ≥ 18 years.
9. Written informed consent that is consistent with ICH-GCP guidelines.

Exclusion Criteria:

1. Prior treatment with EGFR directed small molecules or antibodies.
2. Radiotherapy within 4 weeks prior to randomization, except as follows:

   1. Palliative radiation to target organs other than chest may be allowed up to 2 weeks prior to randomization
   2. Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
3. Active brain metastases (stable for <4 weeks, symptomatic, or leptomeningeal disease). Dexamethasone therapy will be allowed if administered as a stable dose for at least 4 weeks before randomization.
4. Any other current malignancy or malignancy diagnosed within the past three (3) years (other than basal-cell carcinoma of the skin, in situ cervical cancer, in situ prostate cancer).
5. Known pre-existing interstitial lung disease.
6. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g. Crohn's disease, malabsorption or CTC grade >2 diarrhoea of any aetiology, based on investigator assessment.
7. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3 (Refer to Appendix 10.4), unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to randomisation.
8. Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
9. Women of child-bearing potential and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry, for the duration of study participation and for at least 2 months after treatment has ended. Adequate methods of contraception and women of Child-Beanng Potenial are discussed in Section 4.2.2.3.
10. Female patients of childbearing potential (see Section 4.2.2.3) who are nursing or are pregnant.
11. Patients unable to complv with the protocol in the opinion of the investigator.
12. Active hepatitis B infection (detined as presence of Hepatitis B DNA), active hepatitis C infection (defined as vresence of Hepatitis C RNA) and/or known HIV carrier.
13. Known or suspected active drug or alcohol abuse in the opinion of the investigator.
14. Requirement for treatment with any of the prohibited concomitant medications listed in Section 4.2.3.
15. Any contraindications for therapy with gefitinib or erlotinib.
16. Known hypersensitivity to erlotinib, gefitinib or the exipients of any of the trial drugs
17. Major surgery within 4 weeks of starting study treatment.
18. Use of any investigational drug within 4 weeks of randomisation (unless a longer time period is required by local regulations or by the guidelines for the investigational product).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
disease control rate | 2 years

SECONDARY OUTCOMES:
progression free survival | 2 years
adverse events | 2 years
  rash, diarrhea, ILD, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao S, Zhang Z, Fang W, Zhang Y, Zhang Z, Hong S, Ma Y, Zhou T, Yang Y, Huang Y, Zhao H, Zhang L. Efficacy and Tolerability of Erlotinib 100 mg/d vs. Gefitinib 250 mg/d in EGFR-Mutated Advanced Non-small Cell Lung Cancer (E100VG250): An Open-Label, Randomized, Phase 2 Study. Front Oncol. 2020 Nov 10;10:587849. doi: 10.3389/fonc.2020.587849. eCollection 2020. PMID 33244458